CLINICAL TRIAL: NCT05716984
Title: A Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study on the Efficacy and Safety of Recombinant Human Brain Natriuretic Peptide in Improving Type 3 Pulmonary Hypertension.
Brief Title: rhBNP in Type 3 Pulmonary Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, LI ZHAO, professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rhBNP-PH2022
Record Dates: First submitted 2022-09-14; First posted 2023-02-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Group 3 Pulmonary Hypertension
Keywords: rhBNP; Group 3 Pulmonary Hypertension; Right cardiac catheter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recombinant human brain natriuretic peptide (Active Comparator): loading dose 1.5 μg/kg iv, followed by 0.0075 μg/kg·min with micro-pump injection for 72 hours.
  Interventions: Drug: recombinant human brain natriuretic peptide
- placebo (Placebo Comparator): loading dose 1.5 μg/kg iv, followed by 0.0075 μg/kg·min with micro-pump injection for 72 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human brain natriuretic peptide — rhBNP 500μg + 0.9% sodium chloride 50ml, the concentration is 10 μg/ml, loading dose 1.5 μg/kg iv, followed by 0.0075 μg/kg·min with micro-pump injection for 72 hours.
  Arms: recombinant human brain natriuretic peptide
Drug: Placebo — placebo 500μg + 0.9% sodium chloride 50ml, the concentration is 10 μg/ml, loading dose 1.5 μg/kg iv, followed by 0.0075 μg/kg·min with micro-pump injection for 72 hours.
  Arms: placebo

SUMMARY:
Pulmonary hypertension is a common clinical syndrome, which seriously affects the quality of life and survival of patients. Pulmonary hypertension (PH) is defined as an increase in mean pulmonary arterial pressure (mPAP) to ≥20 mmHg at rest as measured invasively by right heart catheterisation (RHC). Pulmonary hypertension can be divided into five types, among which pulmonary hypertension caused by chronic pulmonary diseases and/or hypoxia is called Group 3 pulmonary hypertension, which is the most important factor of pulmonary heart disease. The drugs currently used to treat patients with PAH (prostanoids, endothelin receptor antagonists, phosphodiesterase-5 inhibitors, sGC stimulators) have not been sufficiently investigated in Group 3 PH, except indirect treatment methods such as improving hypoxia and controlling infection.

Recombinant human brain natriuretic peptide (rhBNP) is a biological agent with a molecular weight of 3664Da synthesized by DNA technology. It is availble in China. It has many functions such as diuresis, vasodilation, inhibition of renin-angiotensin-aldosterone and sympathetic nervous systems, etc. RhBNP has been suggested in patients with acute myocardial infarction and congestive heart failure. In view of the dilating effect of rhBNP on pulmonary vessels, it is speculated that rhBNP may reduce type 3 pulmonary hypertension. Based on this hypothesis, we conducted a preliminary clinical trial. The results showed that, compared with the placebo group, after rhBNP was continuously pumped for 24 hours, the pulmonary artery hemodynamic indexes continuously monitored by Swan-Ganz catheter were significantly improved. In view of the pharmacological effect of rhBNP and our previous clinical trial results, this study intends to conduct a prospective, multicenter, placebo-controlled, double-blind clinical trial to evaluate the efficacy and safety of rhBNP in the treatment of patients with group 3 pulmonary hypertension.

DETAILED DESCRIPTION:
The study was divided into three stages, including screening period (3 days), treatment period (72 hours) and follow-up period (10 ± 2 days and 30 ± 5 days). Clinical visits were conducted for 5 times, including admission(screening - V0), V1 (randomization), the end of treatment (V2) and 10 ± 2 days before discharge (V3) in the research center; The telephone interview will be followed up and evaluated on the 30th ± 5 day (V4).

After the subjects signed the informed consent form, they completed all screening tests. The qualified subjects immediately started the basic treatment of Group 3 pulmonary hypertension. Three days later, they underwent right heart echocardiography and Swan-Ganz catheterization. The qualified subjects who met all the inclusion criteria and did not meet all the exclusion criteria were randomly allocated to the rhBNP treatment group or the placebo group at a ratio of 1:1, and the course of treatment was 72 hours. Due to the potential risk of hypotension, blood pressure should be monitored regularly during study drug administration. After the treatment, continue to follow up once by telephone, and the whole study period is 33 ± 5 days. During the whole treatment period, the study doctor recorded symptoms, vital signs, physical examination, and adverse reactions (AE/SAE) according to the requirements of the visit.

Except for emergency safety issues, no protocol violation or exemption is allowed. Therefore, the study must be carried out according to the study design, including the operation items specified in the time and event table.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with acute exacerbation of chronic lung diseases, including: chronic obstructive pulmonary disease, bronchiectasis, obsolete pulmonary tuberculosis, obstructive sleep apnea hypopnea syndrome and thoracic or spinal deformity;
2. At rest, the systolic pressure of pulmonary artery measured by right heart Doppler ultrasound was ≥ 50mmHg;
3. At rest, the mean pulmonary artery pressure (mPAP) measured by Swan Ganz catheter was ≥ 25mmHg with PVR ≥ 3WU and PAWP < 15mmHg;
4. Male or female, age ≥ 18 years old, weight ≥ 30kg ~ ≤ 150kg;
5. WHO fc ≥ II.

Exclusion Criteria:

1. Any other types of pulmonary hypertension;
2. Other active respiratory diseases (such as active pulmonary tuberculosis, pulmonary fibrosis, etc.);
3. Patients requiring invasive mechanical ventilation;
4. At rest, PAWP measured by Swan Ganz catheter was ≥ 15mmhg;
5. Uncontrolled hypertension;
6. Systolic blood pressure < 90mmHg;
7. Dopamine dose ≥ 5 μ g•kg-1•min-1；
8. At rest, Doppler echocardiography confirmed left ventricular outflow tract obstruction or left ventricular systolic dysfunction (EF ≤ 55%);
9. Acute coronary syndrome;
10. Severe renal insufficiency (GFR < 30ml / min / 1.73m2);
11. Significant anemia;
12. Milrinone or levosimendan was used within 30 days before screening;
13. Allergic to any component of rhBNP;
14. Participated in other clinical trials within 30 days before screening;
15. Unable to complete the visit task.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean pulmonary artery pressure (mPAP) | 72 hours
  measured by Swan-Ganz catheter

SECONDARY OUTCOMES:
Systolic pressure of pulmonary artery（PASP） | Day 10±2
  measured by Right heart echocardiography
6MWD | Day 10±2
  6-minute walk distance
WHO fc | 72 hours
  Score Sheet
Oxygen partial pressure | 72 hours
  Arterial blood gas analysis
dyspnea | 72 hours
  Score Sheet
NT-proBNP | 72 hours
  Blood
acute event | Day 30±2
  Symptoms, signs and laboratory examinations

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhao, Doctor, Principal Investigator — Shengjing Hospital
Locations (2):
- China (2):
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frost A, Badesch D, Gibbs JSR, Gopalan D, Khanna D, Manes A, Oudiz R, Satoh T, Torres F, Torbicki A. Diagnosis of pulmonary hypertension. Eur Respir J. 2019 Jan 24;53(1):1801904. doi: 10.1183/13993003.01904-2018. Print 2019 Jan. PMID 30545972
- [Background] Ahmad K, Khangoora V, Nathan SD. Lung Disease-Related Pulmonary Hypertension. Cardiol Clin. 2022 Feb;40(1):77-88. doi: 10.1016/j.ccl.2021.08.005. PMID 34809919
- [Background] Karnati S, Seimetz M, Kleefeldt F, Sonawane A, Madhusudhan T, Bachhuka A, Kosanovic D, Weissmann N, Kruger K, Ergun S. Chronic Obstructive Pulmonary Disease and the Cardiovascular System: Vascular Repair and Regeneration as a Therapeutic Target. Front Cardiovasc Med. 2021 Apr 12;8:649512. doi: 10.3389/fcvm.2021.649512. eCollection 2021. PMID 33912600
- [Background] Pan HY, Zhu JH, Gu Y, Yu XH, Pan M, Niu HY. Comparative effects of recombinant human brain natriuretic peptide and dobutamine on acute decompensated heart failure patients with different blood BNP levels. BMC Cardiovasc Disord. 2014 Mar 4;14:31. doi: 10.1186/1471-2261-14-31. PMID 24593826
- [Background] D'Alto M, Di Marco GM, D'Andrea A, Argiento P, Romeo E, Ferrara F, Lamia B, Ghio S, Rudski LG. Invasive and Noninvasive Evaluation for the Diagnosis of Pulmonary Hypertension: How to Use and How to Combine Them. Heart Fail Clin. 2018 Jul;14(3):353-360. doi: 10.1016/j.hfc.2018.02.010. PMID 29966633
- [Background] Parikh KS, Rajagopal S, Arges K, Ahmad T, Sivak J, Kaul P, Shah SH, Tapson V, Velazquez EJ, Douglas PS, Samad Z. Use of outcome measures in pulmonary hypertension clinical trials. Am Heart J. 2015 Sep;170(3):419-29.e3. doi: 10.1016/j.ahj.2015.06.010. Epub 2015 Jun 19. PMID 26385024